CLINICAL TRIAL: NCT04151095
Title: Examining The Effect of Blood Flow Restricted Aerobic Training on Citrate Synthase Activity in Young Healthy Adults
Brief Title: Examining The Effect of Blood Flow Restricted Aerobic Training on Mitochondrial Adaptations in Young Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brendon Gurd, PhD (Other)
Responsible Party: Sponsor-Investigator, Brendon Gurd, PhD, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BFRT
Record Dates: First submitted 2019-04-02; First posted 2019-11-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Mitochondrial Biogenesis
Keywords: Mitochondria; Exercise training; VO2; Aerobic exercise; Citrate Synthase; Blood flow restriction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation concealment, assessor blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Experimental)
  Interventions: Other: BFR Exercise Training
- CTL (Experimental)
  Interventions: Other: CTL Exercise Training

INTERVENTIONS:
Other: BFR Exercise Training — Participants will complete exercise training on a recumbent bike placed on a 45 degree incline (BFR).
  Arms: BFR
Other: CTL Exercise Training — Participants will complete exercise training on a recumbent bike placed on flat ground (CTL).
  Arms: CTL

SUMMARY:
This parallel-arm trial study investigates the effects of restricting arterial blood flow during cycling exercise on citrate synthase. Participants will be randomized to either a blood flow restricted or non-blood flow restricted exercise training group. Both groups will complete seven, 30-minute exercise sessions over a 14-day period.

ELIGIBILITY:
Inclusion Criteria:

* 3 hours of physical activity per week
* No previous cycling training
* No concurrent involvement in another training program
* Body mass index < 30 kg/m2

Exclusion Criteria:

* Presence of cardiovascular disease
* Presence of metabolic disease
* Taking regular oral medication
* Current smoker

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Citrate Synthase | 3 days prior to start of exercise training and 3 days after completing exercise training
  Fold change in citrate synthase maximal activity

SECONDARY OUTCOMES:
Transcription factor A, mitochondrial (TFAM) | 3 days before training to 3 days after training
  Fold change in TFAM protein
Nuclear respiratory factor, 1 (NRF1) | 3 days before training to 3 days after training
  Fold change in NRF-1 protein
Maximal oxygen consumption (VO2peak) | 3 days before training to 3 days after training
  Change in VO2peak (POST-PRE)
Heart rate (HR) | Every 5 minutes during each of the 7, 30-minute exercise sessions
  Average HR
Revolutions per minute (RPM) | Every 5 minutes during each of the 7, 30-minute exercise sessions
  Average RPM
Blood [lactate] | During all exercise sessions at 10 and 30 minutes
  Average blood lactate concentration
Rating of perceived exertion (RPE) | Every 5 minutes during each of the 7, 30-minute exercise sessions
  Average RPE
Nuclear Factor, Erythroid 2 Like 2 (NFE2L2) | 3 days before training to 3 days after training
  Fold change in NFE2L2
Cytochrome c oxidase (COX) | 3 days before training to 3 days after training
  Fold change in COX
Electromyography (EMG) | Throughout each of the 7, 30-minute exercise sessions
  Median frequency and average amplitude of EMG signal
Near-infrared spectroscopy (NIRS) | Throughout each of the 7, 30-minute exercise sessions
  Deoxygenated hemoglobin and oxygenated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Brendon J Gurd, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Preobrazenski N, Mladen SPS, Causer E, Menezes E, Islam H, Drouin PJ, Tschakovsky ME, Gurd BJ. Mitochondrial and cardiovascular responses to aerobic exercise training in supine and upright positions in healthy young adults: a randomized parallel arm trial. Transl Exerc Biomed. 2025 Mar 26;2(1):9-20. doi: 10.1515/teb-2025-0002. eCollection 2025 May. PMID 40224168